CLINICAL TRIAL: NCT02949414
Title: A Phase I Open-label Study to Assess the Safety, Tolerability and Potential Efficacy of a Novel Tracheal Replacement Consisting of a Tissue-engineered Decellularised Tracheal Scaffold With Seeded Autologous Mesenchymal Cells in Subjects With Severe Tracheal Stenosis or Malacia
Brief Title: A Study to Assess the Safety, Tolerability and Potential Efficacy of a Tracheal Replacement Consisting of a Tissue-engineered Tracheal Scaffold With Seeded Mesenchymal Cells
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Cell Therapy Catapult (Other)
Collaborators: University College, London (Other); Videregen Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-00173-CT2013002
Record Dates: First submitted 2016-01-15; First posted 2016-10-31 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Tracheomalacia; Tracheal Stenosis
Keywords: Malacia; Stenosis; Trachea; Transplant
MeSH Terms: conditions — Tracheomalacia; Tracheal Stenosis; Constriction, Pathologic; Tracheal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tracheal Replacement (Experimental): Each patient will receive surgery to implant the cadaveric decellularised tracheal scaffold seeded with autologous mesenchymal cells and all follow-up procedures.
  Interventions: Procedure: Cadaveric decellularised tracheal scaffold seeded with autologous mesenchymal cells

INTERVENTIONS:
Procedure: Cadaveric decellularised tracheal scaffold seeded with autologous mesenchymal cells — The tracheal graft will be manufactured from cadaveric tracheal scaffold and bone marrow derived mesenchymal cells.

SUMMARY:
This is a phase I study to evaluate the safety, efficacy and tolerability of a novel tracheal replacement therapy using cadaveric de-cellularised tracheal scaffold and patients' own mesenchymal cells isolated from a sample of their bone marrow in patients' who suffer from severe tracheal malacia or stenosis.

DETAILED DESCRIPTION:
This is a phase I study to evaluate the safety, tolerability and potential efficacy of a novel tracheal replacement therapy using a cadaveric tracheal scaffold and patients own mesenchymal cells isolated from a sample of the patients own bone marrow. The study is aimed at treating patients who suffer from severe tracheal stenosis or malacia and for whom conventional therapies are no longer adequate. A total of 4 patients will be treated during the course of this study.

A hospital multi disciplinary team will review the medical history and available treatment options for all potential patients and recommend whether they are suitable for the study. Once patients are approved they will enter an 8 week screening period. During this period bone marrow from the patient will be harvested and the manufacturing of the final graft tissue will start. The manufacturing facility will use a cadaveric donated decellularised tracheal scaffold (supplied by the NHS blood and transplant body) and the patients own cells to make the final investigational product (graft).

The product will be surgically grafted into the patient in place of the damaged tracheal section. The graft will be supported by a stent for the first 6 months with replacements of this stent occurring at week 8 and week 16 post-surgical procedure. Hospitalization for a number of days will be required during this replacement steps. The patient will be followed frequently post surgery to capture any safety and efficacy measures. Long term follow up will continue up to 5 years post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older (all subjects must provide written informed consent)
* Stent or tracheostomy dependent diagnosis of tracheal stenosis or tracheomalacia (Cotton-Myers grade 2 or more)
* Subjects in the above categories for whom further conventional therapies are no longer adequate

Exclusion Criteria:

* Pregnancy
* Subjects unable to provide informed consent
* Prior tracheal transplant
* No viable bone marrow cells within the screening period
* Subjects who have conventional treatment options still available that may have additive impact
* Subject diagnosed or treated for a malignancy within 1 year of study entry or who have previously been diagnosed with a malignancy and have any radiographic or biochemical biomarker evidence of malignancy. Subjects with completely resected basal cell carcinoma or squamous cell carcinoma of the skin or in situ malignancy are not excluded
* Subject with active inflammatory or infectious conditions such as polychondritis, granulomatosis with polyangiitis ('Wegener's'), sarcoidosis or tuberculosis
* Co-morbid moderate or severe chronic obstructive pulmonary disease (COPD) as defined in Global Initiative for COPD, 2011 2, that is unrelated to tracheal stenosis or malacia
* Subjects with known presence of human immunodeficiency virus (HIV) antibody, Hepatitis B surface antigen (HbsAG) or Hepatitis C antibody
* Subject with clinically relevant or recent (within 2 years) history of substance abuse, including alcohol
* Serious medical or psychiatric illness likely to interfere with participation in the study
* Participation in any other clinical trial within previous 30 days of the start of this study or concurrent participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of treatment related SAE's as assessed by CTCAE grades as defined in version 4.0 | Up to 8 months post graft

SECONDARY OUTCOMES:
Efficacy: Post Implant Stent free period | Up to 5 years post implant
Efficacy: Post Implant Tracheostomy free period | Up to 5 years post implant
  Absence of other surgical interventions
Efficacy: Mean Airway Diameter evaluations as captured by CT scans | Up to 5 years post implant
Efficacy: Changes in lung function results using a combination of FEV1, FEF50 and PEFR results | Up to 5 years post implant
Number of treatment related AEs as assessed by CTCAE grading version 4.0 | Upto 5 years post implant

OTHER OUTCOMES:
Changes in Quality of Life assessed using EQ-5D questionnaires | Up to 5 years post graft.
Change in Airway Dyspnoea Voice swallowing Index (ADVS) | Up to 5 years post graft.
Medical Resource Utilisation (MRU) assessed by number and type of tracheal related procedures and treatments post tracheal replacement. | Up to 5 years post graft.
Change in maximum phonation time (MPT) measured in seconds | Up to and including 5 years post graft

CONTACTS AND LOCATIONS:
Overall Officials: Martin Birchall, MD, PhD, Principal Investigator — University College, London
Locations (1):
- Royal Nose Throat and Ear Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study and analysis will be published upon completion.